CLINICAL TRIAL: NCT03398538
Title: A Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Resorbable Glass Fiber Matrix in the Treatment of Diabetic Foot Ulcers
Brief Title: Resorbable Glass Fiber Matrix in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETS Wound Care, LLC (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETS-MG-01
Record Dates: First submitted 2018-01-03; First posted 2018-01-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Foot Ulcer; Ulcer Foot; Diabetic Foot
Keywords: DFU; Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Resorbable Glass Fiber Matrix in the Treatment of Diabetic Foot Ulcers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirragen Wound Matrix Dressing (Experimental): MIRRAGEN™ Advanced Wound Matrix is intended for the use in the management of wounds including diabetic ulcers. Wound matrix dressing to be used per manufacturer instructions for use on diabetic foot wounds in conjunction with offloading and Additional (outer) Dressing Application with moisture retention dressing
  Interventions: Other: Offloading; Other: Additional (outer) Dressing Application; Other: Mirragen Wound Matrix Dressing
- Fibracol Wound Dressing (Active Comparator): A commercially available wound dressing to be used per manufacturer's instructions for use on diabetic foot wounds in conjunction with offloading and Additional (outer) Dressing Application with moisture retention dressing moisture retention dressing
  Interventions: Other: Offloading; Other: Additional (outer) Dressing Application; Other: Fibracol Wound Dressing

INTERVENTIONS:
Other: Offloading — Patient will be offloaded in a diabetic camboot after treatment, or total contact cast if patient cannot be fit with diabetic offloading boot
  Other Names: Pressure relief
Other: Additional (outer) Dressing Application — Application of outer a moisture retentive dressing, and a multi-layer compression dressing.
  Other Names: Outer protective dressing
Other: Mirragen Wound Matrix Dressing — Application of Mirragen to wound site along with standard of care treatment
  Arms: Mirragen Wound Matrix Dressing
Other: Fibracol Wound Dressing — Application of Fibracol Alginate along with standard of care treatment
  Arms: Fibracol Wound Dressing

SUMMARY:
This study is a prospective, multi-center, randomized controlled trial designed to collect patient outcome data on 2 commercially available SOC dressings treatments for Diabetic Foot Wounds

DETAILED DESCRIPTION:
This study is a prospective, multi-center, RCT designed to collect patient outcome data on two commercially available SOC treatments for DFUs. The trial will be single blinded in regard to wound healing assessment (another clinician, other than the investigator at each site will assess wound healing) and confirmation of wound healing will be overseen by an independent adjudication committee made up of wound care experts. The study will last twelve weeks, with a two week screening period prior to enrollment.

There are two standard of care arms in the study:

Arm 1: The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with bioactive resorbable glass fiber dressing, MIRRAGEN™Advanced Wound Matrix, followed by a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

Arm 2: The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with calcium alginate Fibracol dressing followed by a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Presence of a DFU, Wagner 1 (see Appendix B for definitions), extending at least through the dermis provided it is below the medial aspect of the malleolus.
* The index ulcer will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot they must be more than 2 cm distant from the index ulcer.
* Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to SV1 and less than 1-year, as of the date the subject consents for study.
* Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
* Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a Toe Brachial Index (TBI) of > 0.6 is acceptable.
* The target ulcer has been offloaded for at least 14 days prior to randomization.
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* Subject understands and is willing to participate in the clinical study and can comply with weekly visits.

Exclusion Criteria:

* Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
* Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
* Subjects with a history of more than two weeks treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
* Subjects taking a selective COX-2 inhibitor, such as Celecoxib, for any condition.
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
* History of radiation at the ulcer site (regardless of time since last radiation treatment).
* Index ulcer has been previously treated or will need to be treated with any prohibited therapies. (See Section 7.3 of this protocol for a list of prohibited medications and therapies).
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
* Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to randomization. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).
* Subject is pregnant or breast-feeding.
* Presence of diabetes with poor metabolic control as documented with an HbA1c > 12.0 within 90 days of randomization.
* Subjects with end stage renal disease as evidenced by a serum creatinine ≥ 3.0 mg/dL within 6 months of randomization.
* Index ulcer has reduced in area by 20% or more after 14 days of SOC from SV1 to the TV1/randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of index ulcers healed at 12 weeks | 12 weeks
  examine percent of ulcers healed at week twelve

SECONDARY OUTCOMES:
Percentage of index ulcers healed at 6 weeks | 6 week
  examine percent of ulcers healed at week six
Time to heal within 6 and 12 weeks | 6 and 12 weeks
  examine time to healing at both six and twelve weeks
Percent Area Reduction (PAR) at 6 and 12 weeks | 6 and 12 weeks
  examine PAR at both six and twelve weeks
Changes in peripheral neuropathy using Semmes Weinstein Monofilament "10"point discrimination test | 12 weeks
  Each clinical trial participant will be examined by the principal investigator with a Semmes Weinstein monofilament wire at 10 points on the study foot, this standardized exam will be scored out of a total of 10 at each visit and recorded
Changes in wound quality of life, the " Wound Quality of Life Questionnaire" will be given to the clinical trial participants and administered during each visit | 12 weeks
  The Wound-QoL, or wound quality of life questionnaire, measures the disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which are always assessed in retrospect to the preceding seven days. This questionnaire will be given to clinical trial participants at each visit, with the scale scores recorded. Each question is scored. Answers to each item are coded with numbers (0='not at all' to 4='very much'). As noted above the score will be reported with a minimam score of "0" and a maximum score of 68
Change in pain levels during trial, using the FACES pain scales which measure pain on a range of 0-10, zero being no pain and 10 being the most severe pain | 12 weeks
  The FACES pain scale will be administered to the clinical trial participants at each visit. The trial participant will select their pain level with a series of faces that correspond to a number between 0 which implies no pain , up to 10 which implies the most severe pain. The scores will be recorded for each clinical trial participant on each visit
Difference in cellulitis and/or infection at 12 weeks | 12 weeks
  Examine difference in infection rate over twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD, PhD, Principal Investigator — USC / Salsa; Charles M Zelen, DPM, Principal Investigator — Professional Education and Research Institute
Locations (5):
- United States (5):
  - Alan M Jacobs and Associates, St Louis, Missouri
  - Lower Extremity Institute of Research and Therapy, Youngstown, Ohio
  - Martinsville Research Institute, Martinsville, Virginia
  - Professional Education and Research Institute, Roanoke, Virginia
  - Shenandoah Lower Extremity Research Institute, Troutville, Virginia